CLINICAL TRIAL: NCT03672331
Title: International Randomized Study Comparing Personalized, Risk-Stratified to Standard Breast Cancer Screening In Women Aged 40-70
Brief Title: My Personalized Breast Screening
Acronym: MyPeBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UC-0109/1805
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breast Screening
Keywords: standard breast screening - risk-based screening program
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Other): Participants will be screened for breast cancer according to current national/regional guidelines and procedures: with a mammogram and/or tomosynthesis (TS) every 1-3 years starting at age 40-50 years, up to age 69-74 years, with or without ultrasound and MRI depending on breast mammographic density and current recommendations. The national/regional guidelines in use in the including center may be subjected to changes during the study. Guidelines and procedures in the standard arm will be updated accordingly.
  Interventions: Other: Mammogram; Other: Ultrasound; Other: MRI; Other: Tomosynthesis
- Risk-based arm (Experimental): Participants will be screened according to a personalised timetable based on their estimated 5-year risk of developing breast cancer: with a mammography and/or tomosynthesis every 1-4 years with or without ultrasound depending on breast density. Risk estimation will be performed using the following variables: age, family history, previous history of benign breast biopsy, personal hormone and reproductive history, breast mammographic density and genotyping (polygenic risk score). Risk assessment will be conducted using Mammorisk™ for women with at most one first-degree relative with breast or ovarian cancer and using Tyrer-Cuzick™ risk score for those women with more than one first-line first degree relative with breast or ovarian cancer.
  Interventions: Other: Mammogram; Other: Ultrasound; Other: MRI; Other: Tomosynthesis

INTERVENTIONS:
Other: Mammogram — Every 1-4 years according to the national/regional guidelines or personalised schedule according to risk assessment
Other: Ultrasound — As required according to the national/regional guidelines or personalised schedule according to risk assessment
Other: MRI — As required according to the national/regional guidelines or personalised schedule according to risk assessment
Other: Tomosynthesis — As required according to the national/regional guidelines or personalised schedule according to risk assessment

SUMMARY:
MyPeBS is an international randomized, open-label, multicentric, study assessing the effectiveness of a risk-based breast cancer screening strategy (using clinical risk scores and polymorphisms) compared to standard screening (according to the current national guidelines in each participating country) in detecting stage 2 or higher breast cancers.

Women will be differentially screened for 4 years and then, after an end-of-study mammogram, they will return to the routine screening practice. The main study endpoint will be measured at the end of the four years of intervention.

Furthermore, follow up data will be collected for 15 years from study entry for evaluation of long-term cumulative breast cancer incidence and breast cancer-specific survival

ELIGIBILITY:
Inclusion Criteria:

1. Female (whether born female or not)
2. Aged 40 to 70 years old (inclusive)
3. Willing and able to comply with scheduled visits, laboratory tests, and other trial procedures
4. Able to provide written informed consent obtained prior to performing any protocol-related procedures
5. Sufficient understanding of any of the languages used in the study
6. Affiliated to a social security/national healthcare system

Exclusion Criteria:

1. Personal history of breast carcinoma, either invasive or ductal carcinoma in situ (DCIS)
2. Prior history of atypical breast lesion, lobular carcinoma in situ or chest wall irradiation
3. Known condition or suspicion of a very high risk predisposition to breast cancer: germline mutation of BRCA1/2, PALB2, TP53 or equivalent
4. History of bilateral mastectomy
5. Recent abnormal breast finding under work-up (clinically suspect lesion or BI-RADS 4 or 5 image)
6. Psychiatric or other disorders that are not compatible with compliance to the protocol requirements and follow-up
7. Women who do not intend to be followed-up for 4 years

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53142 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of stage 2 and plus breast cancer (non-inferiority analysis) | 4 years
  The study primary objective is to show non-inferiority of the risk-stratified screening strategy in terms of incidence rate of breast cancer of stage 2 and higher (2+), compared to standard screening.

SECONDARY OUTCOMES:
Incidence rate of stage 2 and plus breast cancer (superiority analysis) | 4 years
  The key secondary objective, if non-inferiority is shown, is to demonstrate superiority of the risk-based screening arm to reduce the incidence rate of stage 2+ breast cancer, compared to standard screening.
Rate of morbidity in each arm | 4 years
  Morbidity is defined as false positive imaging findings and benign breast biopsies
Subject anxiety in response to risk evaluation | 4 years
  Subject anxiety will be evaluated using the State-Trait Anxiety Inventory (STAI) questionaire, and compared between treatment arms
Socio-psychological characteristics of subjects | 4 years
  Socio-psychological characteristics will be evaluated using study specific questions concerning comprehension, information-seeking behavior, satisfaction and socio-demographic and economic status
Subject quality of life | 4 years
  Subject quality of life will be evaluated using the EQ-5D quality of life questionnaire
Comparison of cost-effectiveness of each strategy | 4 years
  Crude costs, defined as full real costs per stage 2 cancer diagnosis, will be estimated in each arm. The cost-effectiveness of mammographic screening will be calculated by comparing estimated life-years and costs of breast cancer in each arm
Incidence of stage-specific breast cancer in each arm (including DCIS) | 4 years
  Comparison of the overall incidence of breast cancer detected in each arm according to AJCC stage
Estimates of the rate of detection of clinically non-significant tumours (overdiagnosis) in each study arm | 15 years
  Overdiagnosed breast cancer cases are defined as cancers that would never have been detected clinically, if women had not been screened. Differential overdiagnosis will be measured comparing the cumulative incidence of breast cancer in each arm 15 years after the end of the interventional period of the study.
Rate of false negative images and interval cancers in each arm | 4 years
  False negative images: in case of diagnosis of breast cancer in women whose last screening images (including mammogram +/- US and MRI) were considered as Breast Imaging- Reporting and Data System 1 or 2 (BI-RADS 1 or 2) at 6 months maximum before diagnosis. Interval cancers are defined as a breast cancers diagnosed between a negative screening episode - [mammogram classified as normal (BI-RADS ACR 1 or 2 or equivalent) or abnormal mammogram but negative assessment] and the next planned mammogram
10- and 15-year breast cancer specific survival in MyPeBS and in a combined analysis of the Wisdom and MyPeBS studies | 15 years
Detection rate of stage 2+ breast cancer in women who had screening tomosynthesis (where and when available) and the rate without tomosynthesis | 4 years
Incidence of all stage and stage 2 + breast cancers at 10- and 15-year follow-up | 15 years
Incidence of stage 2 + breast cancer in each arm, in women aged 40-49 at inclusion | 4 years
Rate of breast cancers identified at second reading in each arm | 4 years
Rate of false positive imaging findings and benign breast biopsies in women classified at low risk in risk-based arm | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzette DELALOGE, MD, Study Chair — Gustave Roussy - FRANCE; Paolo GORGIO-ROSSI, MD, Principal Investigator — Arcispedale Santa Maria Nuova-IRCCS - ITALY; Corinne BALLEYGUIER, MD, Principal Investigator — Gustave Roussy - FRANCE; Michal GUINDY, MD, Principal Investigator — ASSUTA Hospital - ISRAEL; Jean-Benoit BURRION, MD, Principal Investigator — Institut Jules Bordet - BELGIUM; Fiona GUILBERT, MD, Principal Investigator — University of Cambridge - UK; Marta ROMÁN, PhD, Principal Investigator — PSMAR - SPAIN
Locations (6):
- Institut Jules Bordet, Brussels, Belgium
- Gustave roussy, Villejuif, France
- Assuta Medical Center Ramat HaHayal, Tel Aviv, Israel
- AUSL Reggio Emilia, Reggio Emilia, Emilia-Romagna, Italy
- Marta Romản, Barcelona, Spain
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
URL: https://www.mypebs.eu/

REFERENCES:
- [Derived] Roux A, Hervouet L, Stefano FD, French DP, Giordano L, Ritchie D, Bugat MR, Keatley D, Cholerton R, McWilliams L, Rossi PG, Balleyguier C, Guindy M, Gilbert FJ, Burrion JB, Roman M, Vissac-Sabatier C, Couch D, Delaloge S, Montgolfier S; MyPeBS Investigators and the MyPeBS Consortium. Acceptability of risk-based breast cancer screening among professionals and healthcare providers from 6 countries contributing to the MyPeBS study. BMC Cancer. 2025 Mar 15;25(1):483. doi: 10.1186/s12885-025-13848-z. PMID 40089664
- [Derived] Roux A, Cholerton R, Sicsic J, Moumjid N, French DP, Giorgi Rossi P, Balleyguier C, Guindy M, Gilbert FJ, Burrion JB, Castells X, Ritchie D, Keatley D, Baron C, Delaloge S, de Montgolfier S. Study protocol comparing the ethical, psychological and socio-economic impact of personalised breast cancer screening to that of standard screening in the "My Personal Breast Screening" (MyPeBS) randomised clinical trial. BMC Cancer. 2022 May 6;22(1):507. doi: 10.1186/s12885-022-09484-6. PMID 35524202
- See also: Public website of MyPeBS — http://www.MyPeBS.eu/